CLINICAL TRIAL: NCT04124744
Title: A Pilot Randomised Controlled Trial of a Volunteer Health Champion Intervention to Support People With Severe Mental Illness to Improve Their Physical Health
Brief Title: A Pilot Randomised Controlled Trial of a Health Champion Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 270290
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Will receive the Health Champion intervention
  Interventions: Other: Health Champions intervention
- Control (Active Comparator): Treatment as usual
  Interventions: Other: Control group-treatment as usual

INTERVENTIONS:
Other: Health Champions intervention — Health Champions are trained volunteers who will support service users with their physical health goals over 9 months, meeting once a week
  Arms: Intervention
Other: Control group-treatment as usual — Participants will receive treatment as usual from their Community Mental Health Team
  Arms: Control

SUMMARY:
This study is a pilot RCT to evaluate the effectiveness and implementation challenges of an intervention using volunteer 'Health Champions' matched with service users to support service their physical health goals.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old with a serious mental illness (Mood [affective] disorders [F30-F39], Schizophrenia, schizotypal, delusional, and other non-mood psychotic disorders [F20-F29]).
* Currently with a Community Mental Health Team (CMHT).
* Want to make changes to their physical health.
* Has capacity to give written informed consent to take part in the project.
* Able to provide a named Care Coordinator or Point of Contact reachable in the event of a health crisis.

Exclusion Criteria:

* • Under 18 years of age

  * Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-02 (Estimated); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
EQ-5D-3L | Change in outcome from baseline at 9 months and 15 months
  Physical health related quality of life measure-The descriptive system element of the EQ-5D questionnaire produces a 5-digit health state profile that represents the level of reported problems on each of the five dimensions of health. A higher score indicates poorer health.
  into a single summary number.

SECONDARY OUTCOMES:
Recovering Quality of Life Questionnaire-ReQOL | Change in outcome from baseline at 9 months and 15 months
  Mental health related quality of life with minimum score of 0 and maximum of 40 The minimum score is 0 and the maximum is 40, where 0 indicates poorest quality of life and 40 indicates the highest quality of life
Patient Activation Measure | Change in outcome from baseline at 9 months and 15 months
  Measure of self management The responses match the respondents to one of four levels of 'activation', each of which reveals insight into a range of health-related characteristics, including behaviours and outcomes.
Multimorbidity Treatment Burden Questionnaire | Change in outcome from baseline at 9 months and 15 months
  Burden of illness with minimum score of 0 and maximum score of 50 with higher score indicating higher burden
De Jong Gierveld Loneliness Scale | Change in outcome from baseline at 9 months and 15 months
  Measure of loneliness. There are negatively (1-3) and positively (4-6) worded items. On the negatively worded items, the neutral and positive answers are scored as "1". Therefore, on questions 1-3 score Yes=1, More or less=1, and No=0. On the positively worded items, the neutral and negative answers are scored as "1". Therefore, on questions 4-6, score Yes=0, More or less=1, and No=1. This gives a possible range of scores from 0 to 6, which can be read as follows:
  (Least lonely) 0 - (Most lonely) 6
Health screenings in last 6 months | change in number of health screenings from baseline at 9 months and 15 months
  Number of health screenings in last 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data for all primary and secondary outcome measures will be made available
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data requests will be reviewed by the team. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Williams J, Fairbairn E, McGrath R, Bakolis I, Healey A, Akpan U, Mdudu I, Gaughran F, Sadler E, Khadjesari Z, Lillywhite K, Sevdalis N. A feasibility hybrid II randomised controlled trial of volunteer 'Health Champions' supporting people with serious mental illness manage their physical health: study protocol. Pilot Feasibility Stud. 2021 May 31;7(1):116. doi: 10.1186/s40814-021-00854-8. PMID 34059148